CLINICAL TRIAL: NCT04356976
Title: Randomised Controlled Trial of Ventralex Hernia Patch Versus Stratafix Suture for Midline Primary Ventral Hernias
Brief Title: Ventralex Vs Stratafix for Primary Ventral Hernias
Acronym: VPatchPriRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VPatchPriRCT
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial comparing Ventralex hernia patch with Stratafix sutures for repair of primary ventral hernias
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the staff responsible for the postoperative care of the patient will be masked for the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ventralex (Experimental): Repair with Ventralex hernia patch in sublay position
  Interventions: Device: Ventralex
- Stratafix (Active Comparator): Repair with Stratafix suture
  Interventions: Other: Stratafix

INTERVENTIONS:
Device: Ventralex — Repair of hernia using Ventralex patch in sublay position
  Arms: Ventralex
Other: Stratafix — Repair of hernia without mesh. Defect closed with Stratafix suture.
  Arms: Stratafix

SUMMARY:
Randomised controlled trial comparing Ventralex Hernia Patch with Stratafix suture for repair of primary ventral hernias in the midline.

DETAILED DESCRIPTION:
Primary hernias in the midline, including umbilical hernias and epigastric hernias, are among the most common conditions requiring surgery.

Mesh-reinforced as well as suture repair are used for the treatment of primary hernias, but for smaller umbilical hernias (diameter 1-3cm), there is little evidence for the superiority of mesh repair. Despite the widely use of composite ventral patch, there are few studies showing the advantage and disadvantage of ventral patch. In recent years, the barbed suture has been widely used in umbilical and incisional hernias, in laparoscopic as well as in open surgery. However, there are no studies comparing ventral patch with slowly absorbable barbed suture in open surgery.

The investigators intend to compare the use of sublay composite mesh (ventral-patch) with non-resorbable barbed prolene suture repair only and investigate recurrence rate and other short and long-term postoperative complications in these two methods.

ELIGIBILITY:
Inclusion Criteria:

* Defect 1-4 cm
* Primary ventral hernia in the midline
* BMI<35

Exclusion Criteria:

* Defect >4cm
* BMI>35
* Recurrent hernia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | One year
  Recurrence diagnosed at clinical and/or radiologic examination

SECONDARY OUTCOMES:
Rate of intra-and postoperative complications | 30 days
  Complications occurring intraoperatively or in the postoperative period
Rate of seroma development | one year
  Seroma confirmed at follow-up examination
Persisting pain | One year
  Postoperative pain rated with the Ventral Hernia Pain Questionnaire. Pain rated on a scale from 1 to 7, with higher scores indicating more severe pain
Mean number of days postoperative sick leave | 30 days
  Postoperative sick leave

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karlskoga Hospital, Karlskoga, Sweden

IPD SHARING:
Plan to Share IPD: No